CLINICAL TRIAL: NCT01009606
Title: Interest for a Relative of Seeing Himself Proposing to Witness Resuscitation of a Family Member Victim of a Cardiac Arrest
Brief Title: Cardiopulmonary Resuscitation Witnessing by a Relative
Acronym: PRESENCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P071239
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-12

CONDITIONS: Cardiac Arrest
Keywords: Out-of-hospital; Emergency; Cardiac arrest; Post-traumatic stress disorder
MeSH Terms: conditions — Heart Arrest; Emergencies; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 : Control : usual strategy (Active Comparator)
  Interventions: Other: Usual strategy
- Arm 2: Comparator : modified strategy (Experimental)
  Interventions: Other: Modified strategy

INTERVENTIONS:
Other: Usual strategy — Usual strategy
  Arms: Arm 1 : Control : usual strategy
Other: Modified strategy — Proposition to a relative to witness the cardiopulmonary resuscitation of a family member and debriefing ot the situation
  Arms: Arm 2: Comparator : modified strategy

SUMMARY:
The bereavement generated by the loss of a family member can induce pathological situations: depressive state, anxiety, post-traumatic stress disorder and complicated grief. These morbid factors can be influenced by the death circumstances and in particular by the possibility given to the family to attend the medical management of the patient. This clinical trial aims to evaluate the psychological consequences of bereavement on the relatives according to the possibility of witnessing the cardiopulmonary resuscitation of a family member. This possibility lies within the scope of a strategy of global management of the relatives.

DETAILED DESCRIPTION:
This clinical trial aims to compare the presence of post-traumatic stress disorder on a relative related to the death of a family member:

Test group: the medical team will propose to the relative to witness the cardiopulmonary resuscitation.

Control group: the medical team will not modify its usual management of care.

ELIGIBILITY:
Inclusion Criteria:

* Patient victim of a cardiac arrest and resuscitation initiated
* Occurrence of cardiac arrest at home
* Presence of a relative :

  * husband or spouse
  * father or mother
  * son or daughter
  * brother or sister
* Patient's age ≥ 18 years
* Relative's age ≥ 18 years
* Consent of the relative to the participation in the study

Exclusion Criteria:

* No understanding of the explanations (language problem, important agitation)
* Non-affiliated to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of relatives having a score of the Impact of Events Scale (IES) > 30 | 3 months

SECONDARY OUTCOMES:
Psychological questionnaires as the hospital anxiety and depression scale (HAD), the Mini International Neuropsychiatric Interview (MINI), the Inventory of Complicated Grief (ICG) | 3 and 12 months
Psychological follow-up | 3 months
Suicide | 3 and 12 months
Medico-legal recourse | 12 months
Quality of the cardiopulmonary resuscitation | day 0
Questionnaire evaluating the stress of the medical and paramedical team | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ADNET, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- SAMU 93 - Hôpital Avicenne, Bobigny, Île-de-France Region, France

REFERENCES:
- [Derived] Jabre P, Bougouin W, Dumas F, Carli P, Antoine C, Jacob L, Dahan B, Beganton F, Empana JP, Marijon E, Karam N, Loupy A, Lefaucheur C, Jost D, Cariou A, Adnet F, Rea TD, Jouven X. Early Identification of Patients With Out-of-Hospital Cardiac Arrest With No Chance of Survival and Consideration for Organ Donation. Ann Intern Med. 2016 Dec 6;165(11):770-778. doi: 10.7326/M16-0402. Epub 2016 Sep 13. PMID 27618681
- [Derived] Jabre P, Tazarourte K, Azoulay E, Borron SW, Belpomme V, Jacob L, Bertrand L, Lapostolle F, Combes X, Galinski M, Pinaud V, Destefano C, Normand D, Beltramini A, Assez N, Vivien B, Vicaut E, Adnet F. Offering the opportunity for family to be present during cardiopulmonary resuscitation: 1-year assessment. Intensive Care Med. 2014 Jul;40(7):981-7. doi: 10.1007/s00134-014-3337-1. Epub 2014 May 23. PMID 24852952
- [Derived] Jabre P, Belpomme V, Azoulay E, Jacob L, Bertrand L, Lapostolle F, Tazarourte K, Bouilleau G, Pinaud V, Broche C, Normand D, Baubet T, Ricard-Hibon A, Istria J, Beltramini A, Alheritiere A, Assez N, Nace L, Vivien B, Turi L, Launay S, Desmaizieres M, Borron SW, Vicaut E, Adnet F. Family presence during cardiopulmonary resuscitation. N Engl J Med. 2013 Mar 14;368(11):1008-18. doi: 10.1056/NEJMoa1203366. PMID 23484827